CLINICAL TRIAL: NCT00846937
Title: Effects of a Plant Stanolester Beverage on Cholesterol Metabolism Among Human Subjects With Ileostoma
Brief Title: Plant Stanol Ester Beverage and Ileostoma Patients
Acronym: STOMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Markku Nissinen/ MD, PhD, Dept. of Medicine, Div. of Gastroenterology
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 3097; U1010G0020
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Ileostoma
Keywords: Cholesterol; Plant stanolester; Beverage; Ileostoma; Serum cholesterol level; serum LDL-cholesterol level; Intestinal cholesterol absorption efficiency
MeSH Terms: interventions — Fatty Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Plant stanolester and fatty acid — Plant stanol ester 2gr/day and fatty acid in a beverage compared to plant stanol ester 2gr /day and placebo

SUMMARY:
We aim to examine efficacy of a plant stanolester beverage to lower serum cholesterol and LDL-cholesterol levels, when given with or without a fatty acid preparation. Study subjects are otherwise healthy proctocolectomized ileostoma patients (n=10), who consume stanolester beverage with or without a fatty acid preparation in a random order for one week period after a standardized low-fat meal. Washout period is 4 weeks. Serum lipids, lipoprotein lipids, sterols and fecal sterols and variables of cholesterol metabolism will be examined accordingly.

ELIGIBILITY:
Inclusion Criteria:

* healthy proctocolectomized subjects with an ileostoma

Exclusion Criteria:

* Chronic illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
serum cholesterol level | After treatment perdiods

CONTACTS AND LOCATIONS:
Overall Officials: Markku J. Nissinen, MD,PhD, Principal Investigator — University of Helsinki; Tatu Miettinen, Professor, Study Director — University of Helsinki
Locations (1):
- University of Helsinki, Department of Medicine, Helsinki, Finland